CLINICAL TRIAL: NCT04489186
Title: Piloting the Clinical Value of Wearable Cardiorespiratory Monitoring for People With Cystic Fibrosis
Brief Title: Continuous Cardiorespiratory Monitoring in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Byteflies (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BF0001
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis
Keywords: wearable; cardiorespiratory monitoring; digital medicine
MeSH Terms: conditions — Cystic Fibrosis | interventions — Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: The study is intended to evaluate the feasibility of a prototype wearable device for continuous cardiorespiratory monitoring in an inpatient and outpatient population with CF in preparation of a larger ambulatory clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All subjects (Experimental): Single arm feasibility study with a wearable device intervention for cardiorespiratory and activity monitoring in subjects with cystic fibrosis.
  Interventions: Device: Wearable device

INTERVENTIONS:
Device: Wearable device — Multimodal electrocardiography (ECG), bioimpedance (bioZ) and tri-axial accelerometry (ACC) monitoring with a single wearable device (Byteflies Sensor Dot) to derive heart rate, respiratory rate and actigraphy.
  Other Names: Byteflies Sensor Dot

SUMMARY:
Cystic Fibrosis (CF) is a disease without a primary cure that requires lifelong care and is characterized by pulmonary exacerbations (PEx). Wearable devices could provide a way for long-term monitoring of disease progression and early signs of PEx to intervene as early as possible, thereby improving long-term outcomes.

This in-hospital feasibility study will assess the ability of Byteflies Sensor Dots to collect relevant cardiorespiratory data in people with CF and its compatibility with clinical workflows, 2) identify candidate digital biomarkers, and 3) collect user feedback from patients and healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Confirmed CF diagnosis as determined by a sweat chloride ≥ 60 mmol/L or the presence of two known disease-causing mutations

Exclusion Criteria:

* Inability to provide written informed consent
* A known allergy to any of the used medical adhesives
* Presence of any type of electronic implanted medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Sensor Dot usability | Up to 24 hours
  Assessed via user (healthcare professional and patient) surveys.
Sensor Dot data quality | Up to 24 hours
  Evaluated by visual examination of recorded electrocardiography (ECG), bioimpedance (bioZ), and accelerometry (ACC) data.

SECONDARY OUTCOMES:
Quality of calculated vital signs: heart rate | Up to 24 hours
  Compare Sensor Dot heart rate (derived from ECG) in beats-per-minute against heart rate as measured by standard hospital equipment.
Quality of calculated vital signs: respiratory rate | Up to 24 hours
  Compare Sensor Dot respiratory rate (derived from bioZ) in breaths-per-minute against respiratory rate as measured by standard hospital equipment.
Cough detection | Up to 24 hours
  Assess if cough events can be derived from the wearable data, as compared to self-reported outcomes.
Screen for candidate digital biomarkers in CF | Up to 24 hours
  Evaluate correlations between the recorded vital sign data (Sensor Dot) and CF severity scores derived from routine pulmonary function testing (PFT, based on Global Lung Function Initiative) and PEx.

CONTACTS AND LOCATIONS:
Overall Officials: Erica A Roesch, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is a device feasibility study. The results will be shared via a publication.